CLINICAL TRIAL: NCT02533882
Title: Dose-Response Effects of Transformative Exercise in Improving Health and Function in Adults With Spinal Cord Injury and Multiple Sclerosis
Brief Title: Lakeshore Examination of Activity and Disability Exercise Response Study
Acronym: LEADERS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Lakeshore Foundation (Other)
Responsible Party: Principal Investigator, James Rimmer, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: F140821001
Record Dates: First submitted 2015-03-06; First posted 2015-08-27 (Estimated); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Multiple Sclerosis; Stroke
MeSH Terms: conditions — Multiple Sclerosis; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Movement to Music (Experimental): The Movement to Music classes are composed of a set of exercises tailored to the specific needs and capabilities of each target group. The class will consist of and aerobic component and a strength component performed to varying music tempos. All movements will be choreographed by qualified dance instructors.
  Interventions: Behavioral: Movement to Music
- Adapted Yoga (Active Comparator): Yoga classes will consist of postures adapted by qualified yoga instructors who have extensive experience in disability.
  Interventions: Behavioral: Adapted Yoga
- Waitlist Control (No Intervention): This group will receive biweekly newsletters on a variety of topics. At the end of this trial, they will receive a home based intervention.

INTERVENTIONS:
Behavioral: Movement to Music
  Arms: Movement to Music
Behavioral: Adapted Yoga
  Arms: Adapted Yoga

SUMMARY:
This study will examine the effectiveness of two types of group exercise classes on the health and functional status in inactive adults age 18-65 with neurological conditions including Multiple Sclerosis, stroke, and spinal cord injury (SCI). Participants will be randomly assigned to one of three groups; Movement to Music, Adapted Yoga, or a waitlist group who will complete a home-based exercise intervention of either Movement to Music or Adapted Yoga.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with stroke
* MS - mild to moderate disability (Patient Determined Disease Steps Score 0-6)
* Able to use arms or arms/legs for exercise
* Ambulatory or use manual wheelchair

Exclusion Criteria:

* Cognitive impairment (Mini-Mental State Exam score < 24)
* Recent weight change (+/- 25 pounds in 1 year)
* Poorly controlled blood pressure
* Cardiovascular disease event within the past six months
* Severe pulmonary disease
* Renal failure
* Current tobacco user or quit within the last six months
* Current use of medications for psychosis
* Active pressure ulcers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2014-12; Primary Completion 2019-07-15 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory Fitness as measured by sub-maximal VO2 | 12 weeks
  Submax VO2 is assessed by the six minute walk test or the six minute push test. Participants wear a portable metabolic cart while walking or pushing
Pain as measured by PROMIS Pain Interference Short Form 8a | 12 weeks
Fatigue as measured by PROMIS Fatigue Short Form 8a | 12 weeks
Loneliness as measured by the Three-Item Loneliness Scale | 12 weeks
Grip Strength as measured by hand grip dynamometer | 12 weeks
Strength as measured by Biodex System 3 Multijoint dynamometer | 12 weeks
  Upper body strength is measured using a closed chain push/pull protocol. Lower body strength is measured using the knee flexion/extension protocol.
Balance as measured by the Timed Up and Go | 12 weeks
  The Timed to Up and Go test is performed using a chair with arms. The participants stand up from the chair, walk to a mark measured three meters from the chair then return back to the seat. A score of greater than or equal to 14 seconds (average) has been shown to indicate a high risk of falling.
Balance as measured by Biodex Limits of Stability | 12 weeks
  The Limits of Stability test is performed on the Biodex SD balance machine using the limits of stability protocol created by Biodex.
Balance as measured by Repeated Chair Stands | 12 weeks
  The repeated chair stands test is performed by asking participants to stand up and sit down 5 times as fast as possible. A score of greater than or equal to 14 seconds (average) has been shown to indicate a high risk of falling.

SECONDARY OUTCOMES:
Health Biomarkers as measured by blood analysis (insulin) | 12 weeks
Health Biomarkers as measured by blood analysis (lipids) | 12 weeks
Health Biomarkers as measured by blood analysis (fasting glucose) | 12 weeks
Blood pressure | 12 weeks
Anthropometric measurements (weight) | 12 weeks
Circumference measurements to be reported as composite ratios (waist circumference, hip circumference, neck circumference) | 12 weeks
Physical Function with Mobility Aid as measured by PROMIS Physical Function with Mobility Aid 455b | 12 weeks
Anxiety as measured by PROMIS Emotional Distress-Anxiety Short Form 8a | 12 weeks
Depression as measured by PROMIS Emotional Distress-Depression Short Form 8a | 12 weeks
Sleep Disturbance as measured by PROMIS Sleep Disturbance Short Form 8a | 12 weeks
Ability to participate in social roles and activities as measured by PROMIS Ability to Participate in Social Roles and Activities Short Form 8a | 12 weeks
Nutrition Self-Efficacy as measured by the Nutrition Self-Efficacy Scale | 12 weeks
Physical Exercise Self-Efficacy as measured by the Physical Exercise Self Efficacy Scale | 12 weeks
PROMIS Pain Intensity Short Form | 12 Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Lakeshore Foundation, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Young HJ, Mehta TS, Herman C, Wang F, Rimmer JH. The Effects of M2M and Adapted Yoga on Physical and Psychosocial Outcomes in People With Multiple Sclerosis. Arch Phys Med Rehabil. 2019 Mar;100(3):391-400. doi: 10.1016/j.apmr.2018.06.032. Epub 2018 Aug 6. PMID 30092206
- [Derived] Rimmer JH, Herman C, Wingo B, Fontaine K, Mehta T. Methodological and clinical implications of a three-in-one Russian doll design for tracking health trajectories and improving health and function through innovative exercise treatments in adults with disability. BMC Med Res Methodol. 2018 Mar 14;18(1):28. doi: 10.1186/s12874-018-0480-3. PMID 29540164